CLINICAL TRIAL: NCT00000293
Title: Effect of Nefazodone on Relapse in Females With Cocaine Abuse
Brief Title: Effect of Nefazodone on Relapse in Females With Cocaine Abuse - 10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-10; P50-09259-10
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — nefazodone

INTERVENTIONS:
Drug: Nefazodone

SUMMARY:
The purpose of this study is to determine the effect of nefazodone on relapse to cocaine use in depressed and non-depressed females with cocaine abuse/dependence.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of nefazodone on relapse to cocaine in women and if a greater effect will be seen in the dependent condition. A relapse and coping skills questionnaire will be utilized to determine the various factors important to the relapse process.

ELIGIBILITY:
Inclusion Criteria:

Female, ages 18-55, cocaine abuse/dependence, use of cocaine 7 days of the last 30 days or of the 30 days prior to current abstinence, less than 90 days current abstinence, at least an 8th grade education.

Exclusion Criteria:

Unstable medical conditions; current use of Hismanal, Seldane, or Propulsid; dx of MR, OBS, bipolar, schizophrenia.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1999-01; Study Completion 2001-12

PRIMARY OUTCOMES:
Retention
Primary drug use
Depression (secondary)
Relapse

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States